CLINICAL TRIAL: NCT06972992
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASC47 Injection, for Subcutaneous Use in Combination With Semaglutide in Participants With Obesity
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASC47 in Combination With Semaglutide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharma (China) Co., Limited (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ASC47-103
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: Chronic Weight Management

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Combo Cohort 1 in participants with obesity (Experimental): Cohort 1, dose 1
  Interventions: Drug: ASC47 +Semaglutide; Drug: Placebo+Semaglutide
- Combo Cohort 2 in participants with obesity (Experimental): Cohort 2, dose 2
  Interventions: Drug: ASC47 +Semaglutide; Drug: Placebo+Semaglutide
- Combo Cohort 3 in participants with obesity (Experimental): Cohort 3, dose 3
  Interventions: Drug: ASC47 +Semaglutide; Drug: Placebo+Semaglutide

INTERVENTIONS:
Drug: ASC47 +Semaglutide — ASC47 single subcutaneous injection + Semaglutide QW for 4 weeks
Drug: Placebo+Semaglutide — Placebo single subcutaneous injection + Semaglutide QW for 4 weeks

SUMMARY:
This will be a phase I, randomized, double-blind, placebo-controlled. This study will be conducted in three periods: the screening period, the treatment period, and the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Subject have provided informed consent before initiation of any study specific procedures
* Females who are not pregnant or breastfeeding, or do not plan to become pregnant within 6 months and are willing to use effective contraceptive measures from the first dose of the investigational product until 3 months after the last dose are eligible.
* No clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and other screening procedures, e.g., Clinical laboratory evaluations (congenital non-hemolytic hyperbilirubinemia as assessed by the Investigator (or sub-I).
* Stable body weight (less than 5% self-reported change within the previous 3 months)

Exclusion Criteria:

* Have obesity traced to a medical cause, suggestive of genetic or syndromic obesity or obesity induced by other endocrinologic disorders, such as hypothyroidism, Cushing syndrome, Prader-Willi syndrome and other conditions.
* Have a history of active or untreated malignancy or are in remission from a clinically significant malignancy (other than basal or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years.
* Have a positive alcohol or drug screen at screening or have a history of alcohol or drug abuse within the past 1 year.
* Have an autoimmune disease, is immunosuppressed or is in any way immunocompromised.
* Have received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month or 5 half-lives of the experimental agent (exception of placebo) prior to the start of the treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2025-04-18 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Adverse events | up to 71 days
  Evaluate the incidence of Serious Adverse Events (SAEs) and Adverse Events (AEs)

SECONDARY OUTCOMES:
Change From Baseline in Body Weight | up to 71 days
  Change from baseline (week 1) to week 10 in body weight was evaluated
Cmax of ASC47 | up to 71 days
  Evaluate the Peak Plasma Concentration of ASC47 in combination with semaglutide.
AUC of ASC47 | up to 71 days
  Evaluate the Area under the plasma concentration versus time curve of ASC47 in combination with semaglutide.
T1/2 of ASC47 | up to 71 days
  Evaluate the Terminal-Phase Half-Life of ASC47 in combination with semaglutide.
CL/F of ASC47 | up to 71 days
  Evaluate the Apparent Systemic Clearance of ASC47 in combination with semaglutide.

CONTACTS AND LOCATIONS:
Locations (1):
- Ascletis Clinical Site, San Antonio, Texas, United States